CLINICAL TRIAL: NCT00606099
Title: A 26 Week Randomized, Open Label, Multi-center Study of the Efficacy and Safety of Telbivudine 600 mg Once Daily Versus Adefovir Dipivoxil 10mg Once Daily in Subjects With Compensated Chronic Hepatitis B and Sub-optimal Response to at Least 48 Weeks of Adefovir Dipivoxil 10 mg
Brief Title: Efficacy and Safety of Telbivudine in Patients With Chronic Hepatitis B
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study was cancelled
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AUS03
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis B
Keywords: Adults; compensated chronic hepatitis B; telbivudin; aedevofir dipivoxil
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir dipivoxil

ARMS (2):
- 1 (Experimental): telbivudine
  Interventions: Drug: telbivudine
- 2 (Active Comparator): adefovir dipivoxil
  Interventions: Drug: adefovir dipivoxil

INTERVENTIONS:
Drug: telbivudine — To compare the rate and pattern of treatment-emergent Hepatitis B virus (HBV) viral genotypic mutations after 24 weeks of treatment.
  Arms: 1
Drug: adefovir dipivoxil — Active Comparator
  Arms: 2

SUMMARY:
This study is designed to evaluate the efficacy and safety of telbivudine 600mg versus adefovir dipivoxil 10mg in patients with compensated chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age.
* Patients with compensated chronic hepatitis B who are currently receiving adefovir 10mg once daily.
* Patients must have received adefovir 10mg once daily for at least 48 weeks continuously and have a sub-optimal response to adefovir therapy (≥4log10 copies of HBV DNA/mL).
* Patient is willing to comply with all study requirements.
* Patient is willing and able to provide written informed consent.

Exclusion Criteria:

* Pregnant or nursing (lactating) women. All women must have a negative pregnancy test at the screening visit.
* Female patients of reproductive potential is unwilling to use double barrier method of contraception (condom plus spermicide or diaphragm plus spermicide).
* Patient is co-infected with hepatitis C virus or HIV.
* Patient has previously taken lamivudine.
* Patient is currently abusing illicit drugs or alcohol.
* Patient is using any investigational drugs or with in the last 30 days.
* Patient is enrolled or plans to enroll in a clinical study involving investigational drug.
* Patient has a history of pancreatitis, hepatic decompsensation, Hepatocellular Carcinoma, or a history of hypersensitivity to telbivudine or adfovir.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Efficacy at 24 weeks of treatment. | 1 yr

SECONDARY OUTCOMES:
To compare biochemical response at week 24 of treatment. To compare changes in viral load at week 24 of treatment. To compare the rate and pattern of treatment-emergent Hepatitis B virus (HBV) viral genotypic mutations after 24 weeks of treatment. | 1yr

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Novartis, Atlanta, Georgia
  - Novartis, Flushing, New York
  - Novartis, Sterling, Virginia